CLINICAL TRIAL: NCT03391843
Title: FOLFOXIRI Combined With Cetuximab as a Neoadjuvant Chemotherapy for EGFR Wild Type Locally Advanced Rectal Cancer:A Phase II Study
Brief Title: Neoadjuvant Chemotherapy Combined With Cetuximab for EGFR Wild Type Locally Advanced Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yeming, Renji Hospital, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018CRC R-002
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Rectal Cancer Stage III
Keywords: Local Advanced Rectal Cancer; Neoadjuvant Chemotherapy; FOLFOXIRI; Cetuximab; EGFR wild type
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI+Cetuximab (Experimental): FOLFOXIRI+Cetuximab regimen:Irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h and cetuximab 500mg/m²,all on day 1 of each 2 weeks cycle for 4-6 cycles.
  Interventions: Drug: FOLFOXIRI+Cetuximab regimen

INTERVENTIONS:
Drug: FOLFOXIRI+Cetuximab regimen — FOLFOXIRI+Cetuximab Irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h +Cetuximab 500mg/m²,all on day 1 of each 2 weeks cycle
  Other Names: CPT 11,CAMPTO，Eloxatin，Xelod，Eloxatin,Erbitux

SUMMARY:
A number of pilot studies had shown high rate of complete resection after neoadjuvant chemotherapy alone for local advanced rectal cancer(LARC), but they did not increase the ratio of pathological complete response (pCR) which was associated with improvement of overall survival (OS). On the other hand,some clinical trials show that triple active cytotoxic agents (Fluorouracil, Oxaliplatin, Irinotecan, FOLFOXIRI) combined with cetuximab for EGFR wild type metastatic colorectal cancer had more effective than double agents.Therefore,a hypothesis is the FOLFOXIRI+Cetuximab as the neoadjuvant chemotherapy regimen might improve the patient's ratio of pCR.

DETAILED DESCRIPTION:
This is a multicenter, phase II trial to assess the efficacy and safety of triplet regimen (FOLFOXIRI) combined with cetuximab for patients with EGFR wild type LARC. After 4 cycles of FOLFOXIRI+cetuximab and 2 weeks later, the patients will be evaluated by senior radiologist, oncologist and surgeon through pelvic MRI, CT and Positron Emission Computed Tomography (PET-CT). The patients will go to surgery (TME) if the tumor response is good enough to have complete resection under the decision of the multidisciplinary team (MDT),otherwise, the patients will receive pelvic radiotherapy(45Grey/25Fraction and 5.4Grey/3Fraction boost to the tumor bed) combined with capecitabine(625 mg/m²,bid po,d1-5,qw), and additional four cycles of modified FOLFOX6 (mFOLFOX6) or Oxaliplatin 135mg/m²plus Capecitabine 1.0/m², bid po(XELOX) of each 3 weeks cycle for 2 cycles chemotherapy before TME. All patients will receive 6-8 cycles of mFOLFOX6 or 4-5 cycles XELOX as adjuvant chemotherapy after TME.

FOLFOXIRI+Cetuximab Irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h + Cetuximab 500 mg/m²,all on day 1 of each 2 weeks cycle for 4-6 cycles,

Other Names:

CPT11，CAMPTO Eloxatin Xelod Erbitux

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to 75 years at diagnosis
2. Diagnosis of rectal adenocarcinoma
3. ECOG status: 0～1
4. Clinical stage II (T3-4, N0) or stage III (T1-4, N1-2)
5. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

1),Leukocytes ≥ 3.0 x109/ L, 2),Absolute neutrophil count (ANC) ≥ 1.5 x109/ L 3),Platelet count ≥ 100 x109/ L, 4),Hemoglobin (Hb) ≥ 9g/ dL. 5),Total bilirubin ≤1.5 x the upper limit of normal (ULN). 6),Alanine aminotransferase (ALT)/Aspartate aminotransferase (AST) ≤ 3 x ULN. 7),Serum creatinine ≤ 1.5 x the ULN. 8),Signed informed consent;

Exclusion Criteria:

1. Patient had received pelvic radiotherapy;
2. Patient had received systemic chemotherapy
3. Pregnant and Nursing women
4. Had metastatic disease
5. Uncontrolled co-morbid illnesses or other concurrent disease
6. Patient had second malignant disease within 5 years
7. Patients refused to signed informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pelvic complete resection rate | Up to 10 weeks
  Pathologic confirmation

SECONDARY OUTCOMES:
The rate of local control | 3 years
  Imaging diagnosis
Disease free survival (DFS) | Three years
  Imaging diagnosis
Overall survival | Three years
  Record document
The rate of receive chemoradiation | Up to 10 weeks
  Record document
The rate of clinical complete response after 4 cycles of FOLFOXIRI | Up to 10 weeks
  Pathologic confirmation
The incidence of >=3 grade adverse events | Two years
  Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ye, Master, Principal Investigator — Department of Radiation Oncology,Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Department of Radiation Oncology,Renji Hospital affiliated to Medical School, Shanghai Jiaotong University, Shanghai, S, China